CLINICAL TRIAL: NCT01236443
Title: A Phase I/II Study of Photodynamic Therapy (PDT) Using 2-[1-hexyloxyethyl]-2-devinylpyropheophorbide-a (HPPH) for the Treatment of High Grade Dysplasia, Carcinoma-in-situ and Early Adenocarcinoma in Barrett's Esophagus
Brief Title: Study of Photodynamic Therapy (PDT) Using HPPH in Barrett's Esophagus
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Roswell Park Cancer Institute (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: RP 00-02
Record Dates: First submitted 2010-11-02; First posted 2010-11-08 (Estimated); Last update posted 2014-01-13 (Estimated); Status verified 2014-01

CONDITIONS: Barrett's Esophagus; CIS; High Grade Dysplasia
MeSH Terms: conditions — Barrett Esophagus | interventions — 2-(1-hexyloxyethyl)-2-devinyl pyropheophorbide-a

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- HPPH (Experimental): 3 mg/m2
  Interventions: Drug: HPPH

INTERVENTIONS:
Drug: HPPH — 3 mg/m2 IV

SUMMARY:
A Study to identify toxicity and optimal photodynamic treatment parameters using the photosensitizer 2-[1-hydroxyethyl]-2-devinylpyropheophorbide-a (HPPH) in high grade dysplasia, carcinoma-in-situ, or early adenocarcinoma in Barrett's esophagus.

ELIGIBILITY:
Inclusion Criteria:

* Patient must have biopsy proven high-grade (severe) dysplasia, carcinoma-in-situ or early stage adenocarcinoma;
* Patient may have received prior therapy; e.g. Nd-YAG laser, radiation therapy or chemotherapy. At least one month must have elapsed between prior treatments and PDT.
* Tumors can be primary or recurrent, Stage 0 or I, N0M (any).
* Patients must have no contraindications to endoscopy.
* Male or female patients must be 18 years old or older. Female patients must not be pregnant and must be practicing a medically acceptable form of birth control or be sterile or post-menopausal. A pregnancy test is required and must be negative.
* Patients must sign an Informed Consent according to FDA guidelines and be acceptable to the RPCI IRB.
* Patients must have a Karnofsky status 50 or above.
* Operable patients are not excluded.

Exclusion Criteria:

* Patients with tumors of grade greater than T-1.
* Porphyria or hypersensitivity to porphyrin or porphyrin-like compounds.
* WBC <2,000; platelet count <50,000, prothrombin time 1.5 times above the upper normal limit.
* Patients with impaired renal and/or hepatic function (total serum bilirubin >3.0 mg/d, serum creatinine >3 mg%, alkaline phosphatase (hepatic) or SGOT >3 times the upper normal limit.
* Patients on concurrent chemotherapy or radiation therapy will be excluded as well as those having received prior treatment for the esophageal cancer within 4 weeks of enrollment.
* If the patient has cancer other than non-melanoma skin cancer they must be deemed disease free by their treating physician.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2000-08; Primary Completion 2003-05 (Actual); Study Completion 2013-04 (Actual)

PRIMARY OUTCOMES:
Toxicity of HPPH at different doses | 2 days

SECONDARY OUTCOMES:
Determine optimal PDT parameters using HPPH in HGD, CIS and Barrett's esophagus | length of study
  Determine optimal PDT parameters using HPPH in HGD, CIS and Barrett's esophagus

CONTACTS AND LOCATIONS:
Overall Officials: Hector Nava, MD, Principal Investigator — Roswell Park Cancer Institute
Locations (1):
- Roswell Park cancer institute, Buffalo, New York, United States